CLINICAL TRIAL: NCT01584960
Title: The Effect of Endurance Training on PSA Doubling Time, Body Composition, Insulin Sensitivity and Inflammation in Patients With Prostate Cancer
Brief Title: The Effect of Endurance Training in Patients With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inge Holm (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Sponsor-Investigator, Inge Holm, Administrator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H-D-2008-015
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Prostate Cancer; Insulin Sensitivity; Body Composition, Beneficial
MeSH Terms: conditions — Prostatic Neoplasms; Insulin Resistance; Glucocorticoid Receptor Deficiency | interventions — Endurance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prostate cancer, endurance training (Experimental): Prostate cancer patients doing 2 years of home-based endurance training Cross over design with a control group with no intervention
  Interventions: Behavioral: endurance training

INTERVENTIONS:
Behavioral: endurance training — 2 years of home-based endurance training

SUMMARY:
The aim of the present study is to investigate the effect of endurance on PSA doubling time in prostate cancer patients with an elevation in PSA following radical prostatectomy for localized cancer. Furthermore, underlying mechanisms such as reduction in inflammatory markers and improvement in insulin sensitivity and body composition are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients with an increase in PSA following radical prostatectomy

Exclusion Criteria:

* severe cardiovascular disease
* severe arthritis
* severe neuropathy
* severe hypertension
* therapy with antidiabetic agents
* other treatment for prostate cancer than radical prostatectomy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
PSA doubling time | 2 years

SECONDARY OUTCOMES:
Insulin sensitivity, body composition and inflammation status | 0 months, 6 months and 24 months of training

CONTACTS AND LOCATIONS:
Overall Officials: Bente K Pedersen, Study Director — Centre of Inflammation and Metabolism, Rigshospitalet
Locations (1):
- Centre of Inflammation and Metabolism, Rigshospitalet, Copenhagen, Copenhagen, Denmark